CLINICAL TRIAL: NCT04970160
Title: Rectovestibular Fistula Which Surgical Approaches?
Acronym: Vestibanus
Status: Completed | Type: Observational
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Magdy, Principle investigator, Aswan University Hospital
Other Study IDs: AswanUH2
Record Dates: First submitted 2021-07-05; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Vestibular Fistulae
Keywords: Vestibular anus,; Anal transposition,; Anorectal malformations; Transfistula anorectoplasty
MeSH Terms: conditions — Anorectal Malformations

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- TSARP: Is a surgical procedure
  Interventions: Procedure: TSARP
- ASARP classic: Surgical procedure
  Interventions: Procedure: Classic ASARP
- PSARP: Surgical procedure
  Interventions: Procedure: PSARP
- Modified ASARP: Surgical procedure
  Interventions: Procedure: Modified ASARP

INTERVENTIONS:
Procedure: TSARP — We make four different surgical operations for female patients with rectovestibular fistula
  Other Names: Transfistula anorectoplasty TFARP
  Groups: TSARP
Procedure: PSARP — Posterior sagittal anorectoplasty
  Other Names: Posterior sagittal anorectoplasty
  Groups: PSARP
Procedure: Classic ASARP — Anterior Sagittal anorectoplasty
  Other Names: Anterior Sagittal anorectoplasty
  Groups: ASARP classic
Procedure: Modified ASARP — External anal sphincter preservation
  Other Names: External anal sphincter preservation
  Groups: Modified ASARP

SUMMARY:
This study was a prospective, randomized, comparative study that included female children with rectovestibular fistulae who were selected from patients with anorectal malformations treated at the pediatric surgical unit, Assiut University Hospital during the period from January 2016 to February 2020. The patients were randomly divided into four groups according to the procedure performed: trans- sphincter anorectoplasty(TSARP), posterior sagittal anorectoplasty, classic anterior sagittal anorectoplasty (ASARP), and modified ASARP.

DETAILED DESCRIPTION:
Background: The management of a vestibular fistula is a challenge for pediatric surgeons. The investigator compared four different operative techniques in terms of postoperative complications, continence, and cosmetic appearance. Patients and methods: This study was a prospective, randomized, comparative study that included female children with rectovestibular fistulae who were selected from patients with anorectal malformations treated at the pediatric surgical unit, Assiut University Hospital during the period from January 2016 to February 2020. The patients were randomly divided into four groups according to the procedure performed: trans- sphincter anorectoplasty(TSARP), posterior sagittal anorectoplasty, classic anterior sagittal anorectoplasty (ASARP), and modified ASARP.

ELIGIBILITY:
Inclusion Criteria:

* Female children aged 6 months to 12 years who had rectovestibular fistulae that had been treated by a single-stage repair were included in this study.

Exclusion Criteria:

* Exclusion criteria were patients with recurrence, previous anorectal surgery.
* Patients with anovestibular fistulae.
* Patients with rectoperineal fistulas.
* Patients with cognitive impairment.

Ages: 6 Months to 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Female children with rectovestibular fistula
Study Population: This study was a randomized, comparative trial involving female children suffering from vestibular fistula taken from among patients with anorectal malformations treated at the pediatric surgical unit, Assiut University Hospital from January 2016 to February 2020. The patients were randomly separated into four groups according to the procedure performed. The different procedures included were TSARP, PSARP, classic ASARP, and modified ASARP. Randomization did by copies the names of the techniques on four separate papers and then the surgeon was blindly chose one paper for each patient. Four pediatric surgeons had experience in ARMs techniques were performed the repair.
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2016-01-01; Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Templeton score | 1 year
  The follow up period is up to one year. scheduled dilatation was followed. Data regarding early (up to 2 weeks) complications, such as wound infection, wound dehiscence, and skin excoriation, and delayed (one months to one year) complications, such as mucosal prolapse, fistula formation, and stenosis, were collected. The anorectal function was measured according to age of continence; younger children who had not attained the age of continence (<3.5 years) had the anocutaneous reflex and anal squeeze on rectal digital examination determined; children older than three and half years had fecal continence rated according to the Templeton score
  . It designates the operative outcome as "good," "fair," or "poor." The scoring performed prospectively during each follow up visit.

SECONDARY OUTCOMES:
Anal continence | 1year
  The assessment period is upto one year. scheduled dilatation was followed. Data regarding early (up to 2 weeks) complications, such as wound infection, wound dehiscence, and skin excoriation, and delayed (one months to one year) complications, such as mucosal prolapse, fistula formation, and stenosis, were collected. The anorectal function was measured according to age of continence; younger children who had not attained the age of continence (<3.5 years) had the anocutaneous reflex and anal squeeze on rectal digital examination determined; children older than three and half years had fecal continence rated according to the Templeton score3
  . It designates the operative outcome as "good," "fair," or "poor." The scoring performed prospectively during each follow up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Abdelmohsen, Principal Investigator — Aswan University

IPD SHARING:
Plan to Share IPD: No